CLINICAL TRIAL: NCT01800240
Title: An Open Label, Randomised, 2-Period, 2-Treatment, 2-Sequence, Crossover, Single-Dose Bioequivalence Study of FDC of Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets 15 mg/850 mg (Test Formulation, Torrent Pharmaceuticals Ltd., India) Versus Actoplus Met® 15 mg/850 mg Tablets (Reference Formulation, Takeda Pharmaceuticals America Inc., USA) in Healthy Human Volunteers Under Fed Conditions.
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd's Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PK-09-182
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Torrent's Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets

SUMMARY:
Objective:

subjects to compare the single dose bioavailability of Torrent's Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets 15 mg/850 mg and Actoplus Met® (pioglitazone hydrochloride and metformin hydrochloride) Tablets 15 mg/850 mg of Takeda Pharmaceuticals America, Inc. USA. Dosing periods of studies were separated by a washout period of 14 days.

Study Design:

Randomized, Two-Way Crossover, Single-Dose, and Open-Label

ELIGIBILITY:
Inclusion Criteria:

The volunteers were included in the study based on the following criteria:

* Sex: male.
* Age: 18 - 45 years.
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

The volunteers were excluded from the study based on the following criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute. Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines,Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics | Pre-dose and 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 14.0, 15.0, 16.0, 17.0, 18.0, 20.0, 24.0, 36.0, 48.0, 72.0, 96.0, 120.0 hours after dose administration.
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd.,, Village Bhat, Gandhinagar, Gujarat, India